CLINICAL TRIAL: NCT07314879
Title: Impact of Interventional Revascularization on the Physiological Assessment of Bystander Coronary Lesions by FFR (ABC-FFR)
Brief Title: Impact of Interventional Revascularization on the Physiological Assessment of Bystander Coronary Lesions by FFR
Acronym: ABC-FFR
Status: Completed | Type: Observational
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: University of Erlangen-Nürnberg Medical School (Other); University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Johannes Michael Altstidl, Physician, Friedrich-Alexander-Universität Erlangen-Nürnberg
Other Study IDs: 12_21 Bc
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
Keywords: Intracoronary Pressure Measurement; Fractional Flow Reserve (FFR); Instantaneous Wave-Free Ratio (iFR); Resting Full-Cycle Ratio (RFR); Chronic Coronary Syndrome (CCS); Cardiology
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Hemodynamic Evaluation of Remote Lesion before & after PCI of Index Lesion — Initial hemodynamic evaluation of the remote, parallel lesion, followed by the planned percutaneous coronary intervention of the index lesion, and a final hemodynamic reevaluation of the remote lesion

SUMMARY:
The ABC-FFR trial examines the understudied hemodynamic interaction between parallel coronary stenoses, as the physiological impact of treating one lesion on the pressure indices of lesions in separate parallel branches is not yet fully understood. This prospective, multicenter study enrolls patients scheduled for percutaneous coronary intervention (PCI) of a designated index lesion who also present with a concurrent remote stenosis in a parallel coronary artery. It evaluates potential changes in fractional flow reserve (FFR) and non-hyperemic pressure ratio (NHPR) measurements within the remote lesion both before and after the index lesion is revascularized.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Scheduled percutaneous coronary intervention for at least one coronary lesion (as indicated by evidence of myocardial ischemia on non-invasive stress imaging, an angiographic stenosis severity >90% diameter stenosis, or an hemodynamically significant intracoronary pressure measurement)
* Additional stenosis of ≥ 30% diameter stenosis in a parallel coronary artery anatomically suitable for wire-based intracoronary pressure assessment

Exclusion Criteria:

* ST-elevation myocardial infarction
* Non-ST-elevation myocardial infarction with immediate invasive strategy recommended by current ESC guidelines (e.g. due to hemodynamic instability, cardiogenic shock, acute heart failure presumed secondary to ongoing myocardial ischemia, recurrent or ongoing chest pain refractory to medical treatment, or life-threatening arrhythmias or cardiac arrest after presentation)
* Acute totally occluded coronary artery
* Unsuitability for intracoronary measurement of FFR (e.g. due to contraindications for the administration of adenosine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were scheduled for percutaneous coronary intervention of at least one coronary index stenosis and had at least one additional remote stenosis in a parallel coronary artery
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
ΔFFR | Baseline
  Difference between fractional flow reserve measurements in the remote lesion after and before percutaneous coronary intervention of the index lesion
Change in Hemodynamic Classification by FFR | Baseline
  Change in hemodynamic classification of the remote lesion with fractional flow reserve after percutaneous coronary intervention of the index lesion

SECONDARY OUTCOMES:
ΔNHPR | Baseline
  Difference between non-hyperemic pressure ratio measurements in the remote lesion after and before percutaneous coronary intervention of the index lesion
Change in Hemodynamic Classification by NHPR | Baseline
  Change in hemodynamic classification of the remote lesion with non-hyperemic pressure ratios after percutaneous coronary intervention of the index lesion

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Steigerwaldklinik Burgebrach, Burgebrach
  - Department of Medicine 1 - Cardiology, Nephrology, Intensive Care and Rhythmology, St. Johannes Hospital Dortmund, Dortmund
  - Deparment of Medicine 2 - Cardiology and Angiology, Friedrich-Alexander-Universität Erlangen-Nürnberg, Erlangen

IPD SHARING:
Plan to Share IPD: No
Privacy and ethical restrictions